CLINICAL TRIAL: NCT05501652
Title: Evaluation of the Safety and Efficacy of a Percutaneously Created Interatrial Shunt in Patients With Chronic Heart Failure Without Pulmonary Vascular Disease
Brief Title: ALLEVIATE-HF-HD Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alleviant Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0005
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ALV1System — The ALV1 system is designed to create a controlled size interatrial shunt via a proprietary intra-cardiac catheter. There is no temporary or permanent implant used to create or maintain the interatrial shunt. The therapy is intended to be delivered in a single procedure administered under general anesthesia in a cardiac catheterization laboratory.

SUMMARY:
Patients with heart failure and reduced left ventricular ejection fraction (HFrEF, EF 25-39%), or mid-range left ventricular ejection fraction (HFmrEF, EF 40-49%), or preserved left ventricular ejection fraction (HFpEF, EF ≥ 50%), with mild to moderate functional limitation will be evaluated for treatment via creation of a no-implant interatrial shunt using clinical, echocardiographic, and invasive hemodynamic data.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA class II if a prior history of > NYHA class II; OR NYHA class III; OR ambulatory NYHA class IV symptoms (paroxysmal nocturnal dyspnea, orthopnea, dyspnea on mild or moderate exertion) at screening visit.
2. Within 12 months of study entry: ≥ 1 HF hospital admission (with HF as the primary or secondary diagnosis); OR treatment with IV diuretics; OR an NT-pro BNP value > 150 pg/ml in normal sinus rhythm, > 450 pg/ml in atrial fibrillation, or a BNP value > 50 pg/ml in normal sinus rhythm, > 150 pg/ml in atrial fibrillation within the past 6 months.
3. Site determined echocardiographic LVEF > 25% as measured by the study specific screening transthoracic echo.
4. Site determined hemodynamic criteria assessed by the screening supine bicycle exercise right heart catheterization test, including each of the components (a)-(b) below:

   a. At rest: i. RAP < 14 mmHg ii. PVR < 3.5 Wood units iii. PAS < 70 mmHg iv. Cardiac Index > 1.9 L/min b. At exercise (25-watts): i. PCWP must have a gradient > 5 mmHg of the RA ii. End-expiratory PCWP ≥ 25 mmHg iii. PVR < 1.8 Wood units [if PVR cannot be obtained (e.g., patient stopped pedaling), TPG < 12 mmHg]

Exclusion Criteria:

1. Presence of advanced heart failure documented in the medical history, defined as one or more of the following:

   1. ACC/AHA/ESC Stage D heart failure, non-ambulatory NYHA Class IV HF
   2. Cardiac index < 2.0 L/min/m2
   3. Inotropic infusion (continuous or intermittent) for EF < 40% within the past 6 months
   4. Patient is on the cardiac transplant waiting list.
2. Presence of uncorrected valve disease documented in the medical history and/or confirmed by the study-specific TTE protocol performed during screening, defined as one or more of the following:

   1. Greater than moderate mitral regurgitation
   2. Greater than moderate mitral stenosis
   3. Greater than mild tricuspid regurgitation
   4. Greater than moderate aortic stenosis
   5. Greater than moderate aortic regurgitation
3. Presence of clinically significant untreated carotid artery stenosis documented in the medical history that is likely to require intervention.
4. Presence of clinically significant un-revascularized coronary artery disease documented in the medical history that is likely to require intervention, defined as epicardial coronary artery stenosis associated with angina or other evidence of coronary ischemia.
5. Presence of hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, cardiac amyloidosis or other infiltrative cardiomyopathy such as hemochromatosis or sarcoidosis.
6. Presence of uncontrolled tachyarrhythmia documented in the medical history.
7. Medical history of one or more of the following cardiac procedures:

   1. MI and/or percutaneous coronary intervention (PCI) within the past 3 months
   2. CABG within the past 3 months
   3. SAVR or TAVR within the past 6 months
   4. MVR or TMVR within the past 6 months
8. Medical history of any implanted pacemaker device.
9. Medical history of cardiac ablation procedure (either for atrial or ventricular arrhythmias) within the past 3 months.
10. Presence of chronic pulmonary disease documented in the medical history, defined by one or more of the following:

    1. Current requirement for continuous home oxygen use
    2. Hospitalization within the past 12 months for treatment of chronic pulmonary disease
    3. Significant chronic pulmonary disease defined as FEV1 < 50% of predicted
    4. If COPD is documented in the medical history and the patient is taking oral or inhaled COPD medication at the time of screening, then a spirometry test is to be performed and patient excluded if FEV1 < 50%.
11. Presence of pulmonary hypertension with PASP ≥ 70 mmHg OR PVR > 3.5 Wood units at rest, documented in the medical history or diagnosed during the initial right heart catheterization.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 1-Month
  The composite incidence of one or more of the following through the 1-month follow-up visit: major adverse cardiac, cerebrovascular and thromboembolic events.
Primary Efficacy Endpoint | 1-Month
  Change in supine exercise PCWP at 25-watts exercise from baseline to Month 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Tbilisi Heart and Vascular, Tbilisi, Georgia

REFERENCES:
- [Derived] Laufer-Perl M, Flint N, Arbel Y, Alenezi F, Kittipibul V, Yaranov D, Shaburishvili T, Amin R, Fudim M. Atrial Mechanics in Heart Failure With Preserved Ejection Fraction: Effect of a No-Implant Interatrial Shunt. Circ Heart Fail. 2025 Oct;18(10):e012573. doi: 10.1161/CIRCHEARTFAILURE.124.012573. Epub 2025 Sep 3. PMID 40899260